CLINICAL TRIAL: NCT06218303
Title: A Clinical Study of a Prototype DAA/TAA Vaccine Targeting MUC1 for Immune Interception and Prevention in Ductal Carcinoma In Situ
Brief Title: Prototype DAA/TAA Vaccine Targeting MUC1 for Immune Interception and Prevention in Ductal Carcinoma In Situ
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Finn, Olivera, PhD (Other)
Collaborators: A Glimmer of Hope Foundation (Unknown); Breast Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Emilia J Diego, MD, Associate Professor of Surgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC 21-208
Record Dates: First submitted 2023-12-29; First posted 2024-01-23 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Ductal Carcinoma in Situ
Keywords: T cells; cancer vaccine; immune checkpoint; lyse tumor cells
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — poly ICLC; Aromatase Inhibitors; Anastrozole; Letrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MUC1 vaccine + adjuvant Hiltonol + Aromatase Inhibitor (Experimental): MUC1 peptide vaccine with poly-ICLC adjuvant Hiltonol administered subcutaneously (SQ) Anastrozole 1 mg, letrozole 2.5 mg, or exemestane 25 mg by mouth daily
  Interventions: Biological: MUC1 Peptide Vaccine; Drug: Hiltonol®; Drug: Aromatase Inhibitor
- Aromatase Inhibitor (Active Comparator): Anastrozole 1 mg, letrozole 2.5 mg, or exemestane 25 mg by mouth daily
  Interventions: Drug: Aromatase Inhibitor

INTERVENTIONS:
Biological: MUC1 Peptide Vaccine — MUC1, a therapeutic vaccine, is a transmembrane glycoprotein and a member of the mucin family of molecules.
  Arms: MUC1 vaccine + adjuvant Hiltonol + Aromatase Inhibitor
Drug: Hiltonol® — A synthetic dsRNA viral mimic and host-defense activator, mimics nature by combining the essential elements of human immunity.
  Other Names: POLY-ICLC
  Arms: MUC1 vaccine + adjuvant Hiltonol + Aromatase Inhibitor
Drug: Aromatase Inhibitor — A type of hormone therapy for cancer used to inhibit aromatase to treat a hormone-related breast cancer.
  Other Names: Anastrozole (Arimidex); Letrozole (Femara); Exemestane (Aromasin)

SUMMARY:
Post-menopausal women with biopsy-proven DCIS will be enrolled into two cohorts. One cohort will receive neoadjuvant therapy with an aromatase inhibitor alone for about 12 weeks prior to surgery at 12 weeks. The second cohort will receive neoadjuvant therapy with an aromatase inhibitor and MUC1 vaccination (MUC1 peptide + Hiltonol®) pre-operatively at baseline, and weeks 2 and 10, followed by surgery at about 12 weeks. Patients in the vaccine cohort will be offered an optional boost vaccine 6 months after surgery.

DETAILED DESCRIPTION:
DCIS is frequently detected by screening mammography, and may develop into invasive disease. However, not all DCIS will progress to invasive breast cancer, and some patients are overtreated. Vaccines for DCIS might facilitate therapeutic de-escalation, and allow less aggressive therapy. The TAA MUC1 is expressed in DCIS, and vaccines specific for MUC1 are safe and decrease the rate of recurrence of high-risk premalignant lesions in colon cancer. This clinical trial is designed to evaluate mechanisms of immune activation and suppression in patients with DCIS, both within the peripheral blood and within the DCIS lesion, and will provide data to guide the development of larger trials to evaluate the impact of a MUC1 vaccine to prevent disease recurrence. Ultimately, vaccine success in intercepting the development of breast cancer will provide critical data for the application of these strategies in breast cancer prevention in high-risk individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal female, 18 years of age or older (no menstrual period for at least 12 months, biochemical menopausal by FSH/LH or S/P oophorectomy)
2. Capable of providing informed consent and willing to comply with study procedures
3. Biopsy-proven ER+ DCIS

   * The signed pathology report from the attending pathologist will be used to determine eligibility
   * Sufficient amount of DCIS remaining in the diagnostic core biopsy block(s) and available for research
   * Patients with DCIS suspicious for microinvasion on core biopsy will be eligible because many of these patients will not have invasion on final pathology
   * Women presenting with concurrent bilateral DCIS are eligible only if both the right and left DCIS lesions are ER+, and tissue from both sides will be analyzed and must meet the criteria below
4. DCIS must be ≥ 1cm based on the extent of calcifications on mammogram, the presence of a mass on ultrasound or enhancement on MRI OR DCIS ≥ 5mm on one single core by pathologic evaluation OR DCIS < 5mm if identified in ≥ 2 cores
5. Candidate for aromatase inhibitor
6. Surgery planned as part of definitive local therapy
7. ECOG PS 0-1
8. Absolute neutrophil count ≥ 1.5 x 109/L
9. Platelet count ≥ 100 x 109/L
10. Hemoglobin ≥ 9 g/dl or ≥ 5.6 mmol/L
11. Creatinine ≤ 1.5X the upper limit of normal OR creatinine clearance ≥ 60 ml/min
12. Total bilirubin ≤ 1.5X the ULN; ≤ 2x ULN for patients with Gilbert's disease
13. AST and ALT ≤ 2.5X ULN
14. INR/PT/aPTT ≤ 1.5X ULN or within the therapeutic range if on anti-coagulation

Exclusion Criteria:

1. Invasive breast cancer > 1mm on pathologic evaluation
2. Second malignancy within the last 5 years (definitively treated superficial non-melanoma skin cancer, melanoma in situ, cervical carcinoma in situ allowed)
3. Current hormone replacement therapy, selective estrogen receptor modulator therapy, or aromatase inhibitor therapy--if yes, wash out of 30 days must occur prior to baseline biopsy for the study
4. Recurrent ipsilateral DCIS
5. Current steroid therapy (doses for physiologic replacement in adrenal dysfunction or for contrast allergy pre-medication for contrast allergy or similar indication allowed, topical, ocular and intranasal steroids allowed)
6. Current Immunomodulator therapy (includes anti-CD20 antibodies)
7. History of autoimmune disease requiring systemic immunosuppression, or active autoimmune disease. Replacement therapy with thyroxine, insulin, and physiologic corticosteroids for adrenal or pituitary insufficiency is acceptable.
8. History of immune deficiency
9. Active infection requiring systemic therapy
10. Any medical or psychiatric condition, substance abuse disorder, medical therapy, or laboratory abnormality that might interfere with the patient's participation for the full duration of the study or compliance with the requirements of the study
11. Known active hepatitis B (hepatitis B surface antigen-reactive) or hepatitis C (hepatitis C virus RNA positive). Patients who are hepatitis B core antibody positive without hepatitis B surface antigen reactivity are eligible. Patients who have antibody for hepatitis C are eligible only if hepatitis C RNA is negative by PCR.
12. Known history of HIV (presence of HIV antibodies for HIV 1 and HIV 2)
13. Received a live vaccine within 30 days of the first dose of treatment
14. History of allergies to any component of the MUC1 vaccine or HiltonolR adjuvant
15. Participation on any investigational vaccine, drug, or device trial within the last 30 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity (of MUC1 vaccine) | At Screening, Week 2, Week 4, Week 6, Week 10, Week 12, Week 16, Week 20, Up to 1 year
  Percentage of patients with a 2-fold or greater increase in serum anti-MUC1 IgG from screening date. Serum IgG is measured using enzyme-linked immunosorbent assay (ELISA).

SECONDARY OUTCOMES:
Adverse Events and Serious Adverse Events Related to Treatment | Up to 2 years
  Number of AEs and SAEs related to study treatment using Common Terminology Criteria for Adverse Events version 5 (CTCAE v.5).
Feasibility (Time to planned surgery) | Up to 2 years
  Percentage of patients who experience a greater than 4-week variation in the time to planned surgery that is related to study participation.

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Diego, MD, Principal Investigator — UPMC Magee Women's Hospital
Locations (1):
- UPMC Magee Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No